CLINICAL TRIAL: NCT05660083
Title: Phase II Trial of Alpelisib With iNOS Inhibitor and Nab-paclitaxel in Patients With HER2 Negative Metastatic or Locally Advanced Metaplastic Breast Cancer (MpBC)
Brief Title: Alpelisib/iNOS Inhibitor/Nab-paclitaxel in Patients With HER2 Negative Metaplastic Breast Cancer (MpBC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMCC-BR22-001
Record Dates: First submitted 2022-10-13; First posted 2022-12-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: HER2-negative Breast Cancer; Metastatic Breast Cancer; Metaplastic Breast Carcinoma; TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — omega-N-Methylarginine; N(6)-(1-iminoethyl)lysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iNOS inhibitor and nab-paclitaxel in combination with alpelisib. (Experimental): iNOS inhibitor and nab-paclitaxel in combination with alpelisib in patients with HER2 negative, metastatic or locally advanced MpBC.
  Interventions: Drug: L-NMMA

INTERVENTIONS:
Drug: L-NMMA — Patients with HER2 negative metastatic or locally advanced MpBC, will receive a combination of an iNOS inhibitor, nab-paclitaxel and alpelisib . As prophylaxis against deep venous thrombosis and hypertension, patients will receive aspirin (81 mg po daily) and amlodipine (10 mg po Days 0-5 each cycle). Metformin will be initiated at 500 mg once daily starting one week prior to treatment to reduce risk of severe hyperglycemia. Based on tolerability and serial blood sugar assessments, metformin dose will be increased to 500 mg twice daily, followed by 500 mg with breakfast and 1000 mg with dinner, followed by further increase to 1000 mg twice daily if needed. Insulin sensitizers and/or SGLT2i will be used as second anti-diabetic agents, if necessary. For prophylaxis of alpelisib rash, patients will be treated with an anti-histamine (cetirizine 10 mg daily) along with alpelisib.
  Other Names: iNOS inhibitor

SUMMARY:
This is a research study to test the safety and effectiveness of using the drug alpelisib together with chemotherapy (nab-paclitaxel) and a drug called L-NMMA in patients with HER2 negative metastatic or locally advanced metaplastic breast cancer, who have not responded to previous treatments.

Participants in this study in addition to the standard care chemotherapy will also receive the drug alpelisib and L-NMMA. The therapies will be administered every 3 weeks (1 cycle) until disease progression, toxicity or until the participant withdraws from the study. The nab-paclitaxel chemotherapy will be administered intravenously on Day 1 of the 3 week cycles. Participants will take the drug alpelisib by mouth once daily at a dose determined by a safety study and the drug L-NMMA will be given intravenously on days 1 to 5 of the 3 week cycles.

DETAILED DESCRIPTION:
This is a Phase II trial with a dose escalation/de-escalation lead-in that will investigate the efficacy and safety of an iNOS inhibitor and nab-paclitaxel in combination with alpelisib in patients with HER2 negative, metastatic or locally advanced MpBC. The prognosis for metastatic or locally advanced metaplastic breast cancer (MpBC), a rare and highly chemotherapy-resistant subtype of TNBC, is even worse than for non-metaplastic TNBC, with a median overall survival ranging from 3 to 8 months.1 Standard systemic chemotherapy remains the only available treatment option for patients with metastatic or locally advanced MpBC, even though this disease is largely refractory to cytotoxic drugs. Therefore, combination strategies to understand and overcome mechanisms of resistance to improve marginal chemotherapeutic efficacy are needed to improve the prognosis of these patients. We have found that inducible nitric oxide synthase (iNOS) is a critical target for overcoming chemotherapy resistance in TNBC.2,3 iNOS expression is increased and associated with poor prognosis in invasive TNBC and MpBC.2-5 It has been shown that nitric oxide (NO) through iNOS induces many of the major oncogenic pathways such as RAS/ERK, HIF1α, NF- κB, and others making this a unique oncogenic driver. One of the major oncogenic pathways activated by iNOS/NO is the phosphatidylinositol 3-kinase (PI3K)/Akt pathway.6-9 Alterations in the Pl3K/Akt pathway have also been linked with chemotherapy resistance, especially in MpBC.10-14 We hypothesize that addition of the PI3K inhibitor, alpelisib, to a pan-NOS inhibitor (L-NMMA) and nab-paclitaxel will increase objective response rate (ORR) in patients with HER2 negative metastatic or locally advanced MpBC. Both first- and second-line patients will be eligible for this trial. Patients may have received prior immunotherapy, per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or legally acceptable representative if applicable) provides written informed consent for the study.
2. At least 18 years of age on the day of informed consent signing.
3. Histologically confirmed HER2 negative MpBC and/or Triple Negative Breast Cancer (TNBC) with squamous and/or sarcomatoid elements, including osseous, chondroid, and spindle morphology.
4. HER2 negative status as defined by the current American Society of Clinical Oncology and College of American Pathologists guidelines at time of study entry.
5. Locally advanced inoperable or metastatic MpBC with measurable disease by RECIST 1.1 Both first- and second-line patients will be eligible for this trial. Patients may have received prior immunotherapy, per standard of care.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Adequate organ and marrow function as defined below:

   * Hemoglobin ≥9.0 g/dl (without blood transfusion within 2 weeks of laboratory test used to determine eligibility)
   * Absolute neutrophil count ≥1000/μL (without granulocyte colony stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
   * Platelet count ≥100,000/μL (without transfusion within 2 weeks of laboratory test used to determine eligibility)
   * Serum total bilirubin (TB) ≤1.5 x institutional upper limit of normal (ULN; In the case of known Gilbert's syndrome, a higher serum TB [>1.5 x ULN] is allowed),
   * Aspartate transaminase/alanine transaminase ≤5 x institutional ULN
   * Creatinine ≤1.5X the ULN or measured creatinine clearance ≥ 60 mL/min/1.
8. Fasting blood glucose of ≤140 mg/dl and HgbA1c ≤7.0.
9. Ability to swallow oral medication.
10. Ability to take aspirin.
11. Women of childbearing potential must agree to use contraception for the duration of the study through 90 days after the last dose of study treatment. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, male participants must not donate sperm during the study and up to the time period as specified in labels of study drugs.
12. If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting the study treatment.
13. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Concomitant use of strong inhibitors or strong inducers of cytochrome P450 (CYP)3A4. The patient must have discontinued strong CYP3A4 inhibitors or strong CYP3A4 inducers for at least 1 week prior to study treatment initiation (Examples included in Appendix 2).
2. Currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis, or otherwise. Therapy with DOACs, heparin, low molecular weight heparin, direct oral anticoagulants or fondaparinux is allowed.
3. Concurrent use of medications that interact with nitrate/nitrite levels (Examples included in Appendix 3).
4. Received previous treatment with nab-paclitaxel, Pl3K inhibitor, AKT inhibitor, or mTOR inhibitor.
5. Known history of Steven Johnson's syndrome or toxic epidermal necrolysis.
6. Since HAART agents are metabolized by CYP3A4, HIV positive patients will be excluded from this trial.
7. Poorly controlled hypertension at baseline (defined as systolic blood pressure >150 mm Hg). Isolated, unconfirmed systolic BP elevations will NOT exclude participation. Patients with medication-controlled hypertension are allowed provided they have been on their current medications for at least 4 weeks prior to Cycle 1, Day 1.
8. Has any of the following cardiac abnormalities:

   * Symptomatic congestive heart failure
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
   * Left ventricular ejection fraction <50% as determined by multigated acquisition scan or echocardiogram
   * Myocardial infarction ~6 months prior to enrollment
   * Unstable angina pectoris
   * Serious uncontrolled cardiac arrhythmia
   * Symptomatic pericarditis
   * History of congenital QT prolongation
   * Absolute corrected QT interval of >480 msec in the presence of potassium >4.0 mEq/L and magnesium >1.8 mg/dl.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks prior to study treatment administration. NOTE: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent.
10. Known or suspected hypersensitivity to any component or excipient of the proposed regimen (nab-paclitaxel, alpelisib, iNOS inhibitor, aspirin).
11. Known additional malignancy that requires active treatment.
12. Pneumonitis/ interstitial lung disease on baseline CT scan of the chest or moderate to severe chronic lung disease
13. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
14. Manifestations of malabsorption due to prior gastrointestinal surgery, gastrointestinal surgery disease, or an unknown reason.
15. Symptomatic/untreated metastatic central nervous system disease.
16. Type I diabetes mellitus irrespective of Hgb A1c OR uncontrolled type II diabetes mellitus defined as hemoglobin A1c >7%.
17. Uncontrolled gastric ulcer
18. ≥ Grade 2 sensory neuropathy
19. Osteonecrosis of jaw
20. Pancreatitis
21. Pregnant, breastfeeding or expecting to conceive children within the projected duration of the study, starting with the prescreening or screening visit through 30 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Define recommended phase II dose (RP2D) | The RP2D will be defined as the highest dose administered at which 6 patients complete treatment with experiencing <2 DLTs (Study completion is an average of 6 cycles, determined by diseases progression, unacceptable toxicity, physician's discretion)
  Define recommended phase II dose (RP2D) of Alpelisib in combination with standard dose of q3wk nab-paclitaxel and L-NMMA
Objective response rate (ORR) | Study treatment will continue until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study. An average of 6 cycles q3week.
  Objective response rate (ORR) of an iNOS inhibitor and nab-paclitaxel in combination with alpelisib in patients with HER2 negative metastatic or locally advanced MpBC.

SECONDARY OUTCOMES:
PFS of patients with HER2 negative metastatic or locally advanced MpBC | Study treatment will continue until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study. An average of 6 cycles q3week.
  Progression-free survival (PFS) of patients with HER2 negative metastatic or locally advanced MpBC treated with an iNOS inhibitor and nab-paclitaxel in combination with alpelisib.
OS of patients with HER2 negative metastatic or locally advanced MpBC | Study treatment will continue until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study. An average of 6 cycles q3week.
  Overall survival (OS) of patients with HER2 negative metastatic or locally advanced MpBC treated with an iNOS inhibitor and nab-paclitaxel in combination with alpelisib.
Analysis of responses to an iNOS inhibitor and nab-paclitaxel in combination with alpelisib. | Study treatment will continue until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study. An average of 6 cycles q3week.
  Analysis of tissue and-blood-based correlates of responses to an iNOS inhibitor and nab-paclitaxel in combination with alpelisib in available specimens.
PIK3CA mutation | Core biopsy will be collected at Baseline and after Cycle 2. Each cycle is 21 days (q3week).
  Tissue will be collected to detect the presence of a PIK3CA mutation (e.g. E545K, E542K, H1047R/Y/L), and efficacy according to PIK3CA mutation status assessed retrospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Polly A Niravath, MD, Principal Investigator — Houston Methodist Cancer Center
Locations (3):
- United States (3):
  - National Institute of Health Clinical Center, Bethesda, Maryland
  - Houston Methodist Neal Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno AC, Lin YH, Bedrosian I, Shen Y, Babiera GV, Shaitelman SF. Outcomes after Treatment of Metaplastic Versus Other Breast Cancer Subtypes. J Cancer. 2020 Jan 1;11(6):1341-1350. doi: 10.7150/jca.40817. eCollection 2020. PMID 32047541
- [Background] Granados-Principal S, Liu Y, Guevara ML, Blanco E, Choi DS, Qian W, Patel T, Rodriguez AA, Cusimano J, Weiss HL, Zhao H, Landis MD, Dave B, Gross SS, Chang JC. Inhibition of iNOS as a novel effective targeted therapy against triple-negative breast cancer. Breast Cancer Res. 2015 Feb 22;17(1):25. doi: 10.1186/s13058-015-0527-x. PMID 25849745
- [Background] Dave B, Gonzalez DD, Liu ZB, Li X, Wong H, Granados S, Ezzedine NE, Sieglaff DH, Ensor JE, Miller KD, Radovich M, KarinaEtrovic A, Gross SS, Elemento O, Mills GB, Gilcrease MZ, Chang JC. Role of RPL39 in Metaplastic Breast Cancer. J Natl Cancer Inst. 2016 Dec 31;109(6):djw292. doi: 10.1093/jnci/djw292. Print 2017 Jun. PMID 28040796
- [Background] Davila-Gonzalez D, Choi DS, Rosato RR, Granados-Principal SM, Kuhn JG, Li WF, Qian W, Chen W, Kozielski AJ, Wong H, Dave B, Chang JC. Pharmacological Inhibition of NOS Activates ASK1/JNK Pathway Augmenting Docetaxel-Mediated Apoptosis in Triple-Negative Breast Cancer. Clin Cancer Res. 2018 Mar 1;24(5):1152-1162. doi: 10.1158/1078-0432.CCR-17-1437. Epub 2018 Jan 4. PMID 29301832
- [Background] Garrido P, Shalaby A, Walsh EM, Keane N, Webber M, Keane MM, Sullivan FJ, Kerin MJ, Callagy G, Ryan AE, Glynn SA. Impact of inducible nitric oxide synthase (iNOS) expression on triple negative breast cancer outcome and activation of EGFR and ERK signaling pathways. Oncotarget. 2017 Jul 26;8(46):80568-80588. doi: 10.18632/oncotarget.19631. eCollection 2017 Oct 6. PMID 29113326
- [Background] Switzer CH, Glynn SA, Cheng RY, Ridnour LA, Green JE, Ambs S, Wink DA. S-nitrosylation of EGFR and Src activates an oncogenic signaling network in human basal-like breast cancer. Mol Cancer Res. 2012 Sep;10(9):1203-15. doi: 10.1158/1541-7786.MCR-12-0124. Epub 2012 Aug 9. PMID 22878588
- [Background] Ridnour LA, Barasch KM, Windhausen AN, Dorsey TH, Lizardo MM, Yfantis HG, Lee DH, Switzer CH, Cheng RY, Heinecke JL, Brueggemann E, Hines HB, Khanna C, Glynn SA, Ambs S, Wink DA. Nitric oxide synthase and breast cancer: role of TIMP-1 in NO-mediated Akt activation. PLoS One. 2012;7(9):e44081. doi: 10.1371/journal.pone.0044081. Epub 2012 Sep 5. PMID 22957045
- [Background] Thomas DD, Ridnour LA, Isenberg JS, Flores-Santana W, Switzer CH, Donzelli S, Hussain P, Vecoli C, Paolocci N, Ambs S, Colton CA, Harris CC, Roberts DD, Wink DA. The chemical biology of nitric oxide: implications in cellular signaling. Free Radic Biol Med. 2008 Jul 1;45(1):18-31. doi: 10.1016/j.freeradbiomed.2008.03.020. Epub 2008 Apr 4. PMID 18439435
- [Background] Prueitt RL, Boersma BJ, Howe TM, Goodman JE, Thomas DD, Ying L, Pfiester CM, Yfantis HG, Cottrell JR, Lee DH, Remaley AT, Hofseth LJ, Wink DA, Ambs S. Inflammation and IGF-I activate the Akt pathway in breast cancer. Int J Cancer. 2007 Feb 15;120(4):796-805. doi: 10.1002/ijc.22336. PMID 17096325
- [Background] Yu HG, Ai YW, Yu LL, Zhou XD, Liu J, Li JH, Xu XM, Liu S, Chen J, Liu F, Qi YL, Deng Q, Cao J, Liu SQ, Luo HS, Yu JP. Phosphoinositide 3-kinase/Akt pathway plays an important role in chemoresistance of gastric cancer cells against etoposide and doxorubicin induced cell death. Int J Cancer. 2008 Jan 15;122(2):433-43. doi: 10.1002/ijc.23049. PMID 17935137
- [Background] Huang WC, Hung MC. Induction of Akt activity by chemotherapy confers acquired resistance. J Formos Med Assoc. 2009 Mar;108(3):180-94. doi: 10.1016/S0929-6646(09)60051-6. PMID 19293033
- [Background] Cai Y, Tan X, Liu J, Shen Y, Wu D, Ren M, Huang P, Yu D. Inhibition of PI3K/Akt/mTOR signaling pathway enhances the sensitivity of the SKOV3/DDP ovarian cancer cell line to cisplatin in vitro. Chin J Cancer Res. 2014 Oct;26(5):564-72. doi: 10.3978/j.issn.1000-9604.2014.08.20. PMID 25400422
- [Background] Li B, Li J, Xu WW, Guan XY, Qin YR, Zhang LY, Law S, Tsao SW, Cheung AL. Suppression of esophageal tumor growth and chemoresistance by directly targeting the PI3K/AKT pathway. Oncotarget. 2014 Nov 30;5(22):11576-87. doi: 10.18632/oncotarget.2596. PMID 25344912
- [Background] Wang Q, Shi YL, Zhou K, Wang LL, Yan ZX, Liu YL, Xu LL, Zhao SW, Chu HL, Shi TT, Ma QH, Bi J. PIK3CA mutations confer resistance to first-line chemotherapy in colorectal cancer. Cell Death Dis. 2018 Jul 3;9(7):739. doi: 10.1038/s41419-018-0776-6. PMID 29970892
- [Background] Takala S, Heikkila P, Nevanlinna H, Blomqvist C, Mattson J. Metaplastic carcinoma of the breast: Prognosis and response to systemic treatment in metastatic disease. Breast J. 2019 May;25(3):418-424. doi: 10.1111/tbj.13234. Epub 2019 Mar 29. PMID 30925636
- [Background] Reddy TP, Rosato RR, Li X, Moulder S, Piwnica-Worms H, Chang JC. A comprehensive overview of metaplastic breast cancer: clinical features and molecular aberrations. Breast Cancer Res. 2020 Nov 4;22(1):121. doi: 10.1186/s13058-020-01353-z. PMID 33148288
- [Background] Somasundaram V, Basudhar D, Bharadwaj G, No JH, Ridnour LA, Cheng RYS, Fujita M, Thomas DD, Anderson SK, McVicar DW, Wink DA. Molecular Mechanisms of Nitric Oxide in Cancer Progression, Signal Transduction, and Metabolism. Antioxid Redox Signal. 2019 Mar 10;30(8):1124-1143. doi: 10.1089/ars.2018.7527. Epub 2018 May 2. PMID 29634348
- [Background] Basudhar D, Bharadwaj G, Somasundaram V, Cheng RYS, Ridnour LA, Fujita M, Lockett SJ, Anderson SK, McVicar DW, Wink DA. Understanding the tumour micro-environment communication network from an NOS2/COX2 perspective. Br J Pharmacol. 2019 Jan;176(2):155-176. doi: 10.1111/bph.14488. Epub 2018 Nov 6. PMID 30152521
- [Background] Janku F, Yap TA, Meric-Bernstam F. Targeting the PI3K pathway in cancer: are we making headway? Nat Rev Clin Oncol. 2018 May;15(5):273-291. doi: 10.1038/nrclinonc.2018.28. Epub 2018 Mar 6. PMID 29508857
- [Background] Cossu-Rocca P, Orru S, Muroni MR, Sanges F, Sotgiu G, Ena S, Pira G, Murgia L, Manca A, Uras MG, Sarobba MG, Urru S, De Miglio MR. Analysis of PIK3CA Mutations and Activation Pathways in Triple Negative Breast Cancer. PLoS One. 2015 Nov 5;10(11):e0141763. doi: 10.1371/journal.pone.0141763. eCollection 2015. PMID 26540293
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Background] Kriegsmann M, Endris V, Wolf T, Pfarr N, Stenzinger A, Loibl S, Denkert C, Schneeweiss A, Budczies J, Sinn P, Weichert W. Mutational profiles in triple-negative breast cancer defined by ultradeep multigene sequencing show high rates of PI3K pathway alterations and clinically relevant entity subgroup specific differences. Oncotarget. 2014 Oct 30;5(20):9952-65. doi: 10.18632/oncotarget.2481. PMID 25296970
- [Background] Zhai J, Giannini G, Ewalt MD, Zhang EY, Invernizzi M, Niland J, Lai LL. Molecular characterization of metaplastic breast carcinoma via next-generation sequencing. Hum Pathol. 2019 Apr;86:85-92. doi: 10.1016/j.humpath.2018.11.023. Epub 2018 Dec 8. PMID 30537493
- [Background] Hennessy BT, Gonzalez-Angulo AM, Stemke-Hale K, Gilcrease MZ, Krishnamurthy S, Lee JS, Fridlyand J, Sahin A, Agarwal R, Joy C, Liu W, Stivers D, Baggerly K, Carey M, Lluch A, Monteagudo C, He X, Weigman V, Fan C, Palazzo J, Hortobagyi GN, Nolden LK, Wang NJ, Valero V, Gray JW, Perou CM, Mills GB. Characterization of a naturally occurring breast cancer subset enriched in epithelial-to-mesenchymal transition and stem cell characteristics. Cancer Res. 2009 May 15;69(10):4116-24. doi: 10.1158/0008-5472.CAN-08-3441. Epub 2009 May 12. PMID 19435916
- [Background] Afkhami M, Schmolze D, Yost SE, Frankel PH, Dagis A, Amanam IU, Telatar M, Nguyen K, Yu KW, Luu T, Pillai R, Aoun PA, Mortimer J, Yuan Y. Mutation and immune profiling of metaplastic breast cancer: Correlation with survival. PLoS One. 2019 Nov 6;14(11):e0224726. doi: 10.1371/journal.pone.0224726. eCollection 2019. PMID 31693690
- [Background] Chan JJ, Tan TJY, Dent RA. Novel therapeutic avenues in triple-negative breast cancer: PI3K/AKT inhibition, androgen receptor blockade, and beyond. Ther Adv Med Oncol. 2019 Oct 9;11:1758835919880429. doi: 10.1177/1758835919880429. eCollection 2019. PMID 31636720
- [Background] Andre F, Ciruelos E, Rubovszky G, Campone M, Loibl S, Rugo HS, Iwata H, Conte P, Mayer IA, Kaufman B, Yamashita T, Lu YS, Inoue K, Takahashi M, Papai Z, Longin AS, Mills D, Wilke C, Hirawat S, Juric D; SOLAR-1 Study Group. Alpelisib for PIK3CA-Mutated, Hormone Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2019 May 16;380(20):1929-1940. doi: 10.1056/NEJMoa1813904. PMID 31091374
- [Background] Reddy T, et al. Combination PI3K and NOS targeted therapy for metaplastic breast cancer (abstract). In: European Journal of Cancer, Molecular Targeted Agents. 2020; 138:S49-S50.
- [Background] Nelson RA, Guye ML, Luu T, Lai LL. Survival outcomes of metaplastic breast cancer patients: results from a US population-based analysis. Ann Surg Oncol. 2015 Jan;22(1):24-31. doi: 10.1245/s10434-014-3890-4. Epub 2014 Jul 11. PMID 25012264
- [Background] Rayson D, Adjei AA, Suman VJ, Wold LE, Ingle JN. Metaplastic breast cancer: prognosis and response to systemic therapy. Ann Oncol. 1999 Apr;10(4):413-9. doi: 10.1023/a:1008329910362. PMID 10370783
- [Background] Moulder S, Helgason T, Janku F, Wheler J, Moroney J, Booser D, Albarracin C, Morrow PK, Atkins J, Koenig K, Gilcrease M, Kurzrock R. Inhibition of the phosphoinositide 3-kinase pathway for the treatment of patients with metastatic metaplastic breast cancer. Ann Oncol. 2015 Jul;26(7):1346-52. doi: 10.1093/annonc/mdv163. Epub 2015 Apr 15. PMID 25878190